CLINICAL TRIAL: NCT01304082
Title: A Single-center, Randomized, Double-blind Clinical Study to Evaluate the Effect of pH on Pain Upon Local Anesthetic Administration.
Brief Title: Clinical Study to Evaluate the Effect of pH on Pain Upon Local Anesthetic Administration.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian Wainger, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010-P-000533
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Local Anesthetics
Keywords: pain pH local anesthetics
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline
- lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine
- alkalinized lidocaine (Experimental)
  Interventions: Drug: alkalinized lidocaine

INTERVENTIONS:
Drug: Lidocaine — 1 ml subcutaneous injection of 0.9% lidocaine, given once
  Arms: lidocaine
Drug: normal saline — 1 ml subcutaneous injection 0.9% sodium chloride, given once
  Arms: normal saline
Drug: alkalinized lidocaine — 1 ml subcutaneous injection of 0.9% lidocaine and 0.84% sodium bicarbonate
  Arms: alkalinized lidocaine

SUMMARY:
When one receives a local anesthetic, such as novocaine for a dental procedure, there is a burning painful sensation experienced upon injection of the local anesthetic. We are trying to understand the role of pH (how acidic a solution is) in the production of pain during local anesthetic administration. We hypothesize that less acidic solutions produce less burning. We also want to determine whether or not the pH of the solution affects the rate of onset of the local anesthesia. We will recruit subjects from patients who have a clinical indication for lumbar medial branch (LMB) nerve blocks, procedures frequently performed at the Massachusetts General Hospital Center for Pain Medicine. For each patient, three nerve blocks are administered at adjacent spinal levels, typically using either lidocaine or bicarbonate-buffered lidocaine as the local anesthetic. We will add a saline control as part of the research procedure and then provide lidocaine at the control location before continuing with the nerve blocks. This clinical procedure offers an ideal opportunity to compare the effects of the three solutions. There will be almost no deviation from the standard clinical procedure. After the injection of each solution, the pain score on administration of the medication will be recorded immediately. We will also provide a continuous stimulation (pin taps) after the local anesthetic injection and record when the patient experiences hypoesthesia (reduced sensation) and anesthesia (absent sensation). Finally, we will record the pain score upon reinsertion of a needle to mark the precise location (part of the clinical procedure) one minute after the local anesthetic injection. All data will be collected during the a single clinical visit.

The study will conclude when 60 subjects have successfully been tested. Data will be reviewed annually.

ELIGIBILITY:
Inclusion Criteria:

* patients at MGH Center for Pain Medicine who have clinical indication for undergoing diagnostic medial branch block of nerves to facet joints.

Exclusion Criteria:

* contraindication to the clinical procedure
* do not speak English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Wainger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- C, L, A: control, lidocaine, alkalinized lidocaine
- C, A, L: control, alkalinized lidocaine, lidocaine
- L, C, A: lidocaine, control, alkalinized lidocaine
- A, C, L: alkalinized lidocaine, control, lidocaine
- A, L, C: alkalinized lidocaine, lidocaine, control
Period: Overall Study
Arm/Group | C, L, A | C, A, L | L, C, A | A, C, L | A, L, C
Started | 3 | 2 | 11 | 8 | 5
First Intervention | 3 | 2 | 11 | 8 | 5
Second Intervention | 3 | 2 | 11 | 8 | 5
Third Intervention | 3 | 2 | 11 | 8 | 5
Completed | 3 | 2 | 11 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: One participant was missing age.
  years
    number analyzed (Participants) | 28
    (all) | 54.5 [44.5 to 62.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Baseline Pain Score [Median (Inter-Quartile Range); unit: units on a scale] — This pain score is a validated 11-point numeric rating scale in which patients rate pain between 0 (no pain) and 10 (worst pain imaginable).
  units on a scale | 6 [4 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Rank-transformed Pain Score
Description: Pain score upon injection of local anesthetic:
  the pain score is a validated 11-point numeric rating scale in which patients rate pain between 0 (no pain) and 10 (worst pain imaginable).
Time Frame: immediate, upon injection of each solution
Measure: Least Squares Mean (95% Confidence Interval); unit: rank
Arm/Group | Normal Saline | Lidocaine | Alkalinized Lidocaine
Number analyzed (Participants) | 29 | 29 | 29
rank
  Rank-transformed pain score | 1.97 [1.62 to 2.31] | 2.10 [1.76 to 2.45] | 1.93 [1.59 to 2.27]
  Difference compared to control | 0 [0 to 0] | 0.138 [-0.459 to 0.735] | -0.034 [-0.632 to 0.563]
  Difference compared to lidocaine | -0.138 [-0.735 to 0.459] | 0 [0 to 0] | -0.172 [-0.769 to 0.425]
Statistical Analysis 1: Comparison: Normal Saline vs Lidocaine vs Alkalinized Lidocaine; Analysis: Non-parametric Friedman ANOVA test on rank-transformed outcome with Bonferroni correction for pairwise comparisons. Null hypothesis: No difference between the groups; Test type: Superiority or Other; p = 0.7535, non-parametric Friedman ANOVA test — Bonferroni correction for pairwise comparisons

2. Secondary Outcome: Rank-transformed Time (Seconds) Until Hypoesthesia
Description: Rank-transformed time (seconds) until hypoesthesia will be assessed using a sensory stimulus
Time Frame: 0-180 seconds after each injection.
Measure: Least Squares Mean (95% Confidence Interval); unit: rank
Arm/Group | Normal Saline | Lidocaine | Alkalinized Lidocaine
Number analyzed (Participants) | 29 | 29 | 29
rank
  Rank-transformed time (s) | 2.95 [2.75 to 3.15] | 1.47 [1.27 to 1.67] | 1.59 [1.39 to 1.79]
  Difference compared to control | 0 [0 to 0] | -1.48 [-1.83 to -1.13] | -1.36 [-1.71 to -1.01]
  Difference compared to lidocaine | 1.48 [1.13 to 1.83] | 0 [0 to 0] | 0.121 [-0.228 to 0.469]
Statistical Analysis 1: Comparison: Normal Saline vs Lidocaine vs Alkalinized Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, non-parametric Friedman ANOVA test — Bonferroni correction for pairwise comparisons

3. Secondary Outcome: Rank-transformed Time (Seconds) Until Anesthesia
Description: Rank-transformed time (seconds) until anesthesia will be assessed using a repeated sensory stimulus.
Time Frame: 0-180 seconds after each injection
Measure: Least Squares Mean (95% Confidence Interval); unit: rank
Arm/Group | Normal Saline | Lidocaine | Alkalinized Lidocaine
Number analyzed (Participants) | 29 | 29 | 29
rank
  Rank-transformed time (s) | 2.90 [2.68 to 3.11] | 1.62 [1.40 to 1.84] | 1.48 [1.26 to 1.70]
  Difference compared to control | 0 [0 to 0] | -1.28 [-1.66 to -0.90] | -1.41 [-1.79 to -1.03]
  Difference compared to lidocaine | 1.28 [0.90 to 1.66] | 0 [0 to 0] | -0.14 [-0.52 to 0.24]
Statistical Analysis 1: Comparison: Normal Saline vs Lidocaine vs Alkalinized Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, non-parametric Friedman ANOVA test — Bonferroni correction for pairwise comparisons

4. Secondary Outcome: Rank-transformed Pain Score Upon Needle Stick.
Description: Pain score upon needle stick:
  The pain score is a validated 11-point numeric rating scale in which patients rate pain between 0 (no pain) and 10 (worst pain imaginable).
Time Frame: 1 minute after each injection
Measure: Least Squares Mean (95% Confidence Interval); unit: rank
Arm/Group | Normal Saline | Lidocaine | Alkalinized Lidocaine
Number analyzed (Participants) | 29 | 29 | 29
rank
  Rank-transformed pain score | 2.72 [2.50 to 2.95] | 1.64 [1.41 to 1.86] | 1.64 [1.41 to 1.86]
  Difference compared to control | 0 [0 to 0] | -1.09 [-1.48 to -0.70] | -1.09 [-1.48 to -0.70]
  Difference compared to lidocaine | 1.09 [0.70 to 1.48] | 0 [0 to 0] | 0 [-0.39 to 0.39]
Statistical Analysis 1: Comparison: Normal Saline vs Lidocaine vs Alkalinized Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, non-parametric Friedman ANOVA test — Bonferroni correction for pairwise comparisons

ADVERSE EVENTS:
Arm/Group | Normal Saline | Lidocaine | Alkalinized Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No